CLINICAL TRIAL: NCT02174471
Title: REgression in Left Ventricular Interstitial Expansion and Fibrosis After Aortic Stenosis Surgery
Brief Title: Regression of Myocardial Fibrosis After Aortic Valve Replacement
Acronym: RELIEF-AS
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: ReDA ID 07/0166
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis; Aortic Valve Replacement; T1 Mapping; Extracellular Volume Fraction; Cardiovascular Magnetic Resonance; Diffuse Myocardial Fibrosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Plasma; myocardial biopsy obtained intra-operatively.
Oversight: Data Monitoring Committee: No

SUMMARY:
Aortic stenosis (AS) is the most common valvular heart condition in the United Kingdom and the Western world. Surgery for severe AS prior to symptom onset is controversial. Conventionally changes in valve area and gradient are used to time intervention but myocardial changes may be more predictive of surgical need.

This study aims to elucidate the role of diffuse myocardial fibrosis as a prognostic marker, implementing a novel, non-invasive MRI technique to measure it.

Design: The investigators will measure diffuse myocardial fibrosis in 150 patients with severe narrowing of the aortic valve before and one year after valve replacement. Expected outcomes: Diffuse myocardial fibrosis measured by MRI scanning will predict outcome after surgery in aortic stenosis. Anticipated Health Benefits: Identify patients with higher post operative morbidity and mortality, who may benefit from earlier valve replacement.

DETAILED DESCRIPTION:
Surgery for severe aortic stenosis (AS) prior to symptom onset is controversial. Conventionally changes in valve area and gradient are used to time intervention but myocardial changes may be more predictive of surgical need. This study aims to elucidate the role of diffuse myocardial fibrosis as a prognostic marker, implementing a novel, non-invasive technique to measure it.

AS is the most common valvular heart condition in the United Kingdom and the Western world. Its prevalence rises with age - about 3% aged over 75 have severe AS. During a period of progressive valve narrowing, the left ventricle (LV) adapts to the increased pressure with increasing concentric muscle hypertrophy. However, eventually this remodelling becomes maladaptive and the LV less compliant, leading to symptoms (breathlessness, chest pain, and loss of consciousness). This heralds a significant increase in morbidity and mortality. Consequently aortic valve replacement (AVR) in symptomatic patients is a Class I indication. In most asymptomatic patients however, prophylactic surgery is controversial: the risk of surgery is thought to be greater than watchful waiting, although there is no randomised data to support this approach. Conversely, diffuse myocardial fibrosis is thought to play a key role in functional deterioration, symptom development and possibly outcome in AS. Unfortunately, assessment of AS severity, including hemodynamic parameters such as peak velocity and mean gradient, poorly predict symptom development and/or optimal timing of surgery.

A non-invasive technique to quantify diffuse myocardial fibrosis against the gold standard of myocardial biopsy has been developed and validated in patients with AS: Cardiovascular magnetic resonance (CMR) with T1 mapping uses the extracellular tracer gadolinium to measure the extracellular volume (ECV), which closely reflects the degree of diffuse fibrosis. An important observation in a previous cohort (Flett et al European Heart Journal Cardiovascular Imaging 2012) was the fate of patients with severe fibrosis: they were more symptomatic at baseline, improved the most post-operatively and yet carried a trend towards increased mortality at six months. To unravel this, this study aims to track diffuse fibrosis in the RELIEF-AS study with a larger cohort (n=150) and for longer (12 months) to understand how to use diffuse fibrosis as a prognostic marker.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis (1 or more of: aortic valve area < 1.0cm2, peak pressure gradient >64mmHg, or mean pressure gradient > 40mmHg).
* Symptomatic.
* Age > 18 years and < 90 years.

Exclusion Criteria:

* Severe valvular disease other than AS.
* Previous Valve surgery
* Severe renal impairment eGFR < 30ml/min.
* Any absolute contraindication to CMR
* Other medical condition that limits life expectancy or precludes AVR.
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic stenosis awaiting valve replacement recruited from cardiology outpatient department or as cardiology inpatients.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death | 12 months
Major adverse cardiovascular events (MACE) | 12 months
  MACE: hospitalisation with heart failure, chest pain, syncope, arrhythmia or stroke

SECONDARY OUTCOMES:
Functional improvement | 12 months
  Improvement in 6 minute walk test.
Regression of diffuse myocardial fibrosis | 12 months
  Diffuse myocardial fibrosis measured by T1 mapping by CMR

OTHER OUTCOMES:
LV remodeling post AVR | 12 months
  LV remodeling post AVR measured by CMR and transthoracic echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: James C Moon, MD, Principal Investigator — University College, London
Locations (1):
- The Heart Hospital, University College London Hospitals, London, United Kingdom

REFERENCES:
- [Background] Flett AS, Hayward MP, Ashworth MT, Hansen MS, Taylor AM, Elliott PM, McGregor C, Moon JC. Equilibrium contrast cardiovascular magnetic resonance for the measurement of diffuse myocardial fibrosis: preliminary validation in humans. Circulation. 2010 Jul 13;122(2):138-44. doi: 10.1161/CIRCULATIONAHA.109.930636. Epub 2010 Jun 28. PMID 20585010
- [Background] Flett AS, Sado DM, Quarta G, Mirabel M, Pellerin D, Herrey AS, Hausenloy DJ, Ariti C, Yap J, Kolvekar S, Taylor AM, Moon JC. Diffuse myocardial fibrosis in severe aortic stenosis: an equilibrium contrast cardiovascular magnetic resonance study. Eur Heart J Cardiovasc Imaging. 2012 Oct;13(10):819-26. doi: 10.1093/ehjci/jes102. Epub 2012 May 25. PMID 22634740
- [Derived] Bhuva AN, Treibel TA, De Marvao A, Biffi C, Dawes TJW, Doumou G, Bai W, Patel K, Boubertakh R, Rueckert D, O'Regan DP, Hughes AD, Moon JC, Manisty CH. Sex and regional differences in myocardial plasticity in aortic stenosis are revealed by 3D model machine learning. Eur Heart J Cardiovasc Imaging. 2020 Apr 1;21(4):417-427. doi: 10.1093/ehjci/jez166. PMID 31280289
- [Derived] Smith A, Moravcova S, Treibel TA, Colque-Navarro P, Mollby R, Moon JC, Hamilton-Davies C. Relationship between endotoxin core, staphylococcal and varicella antibody levels and outcome following aortic valve replacement surgery: a prospective observational study. Perioper Med (Lond). 2018 Sep 20;7:20. doi: 10.1186/s13741-018-0101-z. eCollection 2018. PMID 30250733
- [Derived] Treibel TA, Kozor R, Schofield R, Benedetti G, Fontana M, Bhuva AN, Sheikh A, Lopez B, Gonzalez A, Manisty C, Lloyd G, Kellman P, Diez J, Moon JC. Reverse Myocardial Remodeling Following Valve Replacement in Patients With Aortic Stenosis. J Am Coll Cardiol. 2018 Feb 27;71(8):860-871. doi: 10.1016/j.jacc.2017.12.035. PMID 29471937
- [Derived] Treibel TA, Kozor R, Fontana M, Torlasco C, Reant P, Badiani S, Espinoza M, Yap J, Diez J, Hughes AD, Lloyd G, Moon JC. Sex Dimorphism in the Myocardial Response to Aortic Stenosis. JACC Cardiovasc Imaging. 2018 Jul;11(7):962-973. doi: 10.1016/j.jcmg.2017.08.025. Epub 2017 Nov 15. PMID 29153564